CLINICAL TRIAL: NCT04540861
Title: Managed Access Program (MAP) to Provide Access to Siponimod Treatment for Patients Diagnosed With Secondary Progressive Multiple Sclerosis With no Satisfactory Alternative Treatment
Brief Title: Managed Access Program (MAP) for Patients Diagnosed With Secondary Progressive Multiple Sclerosis With Active Disease
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBAF312A2001M
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: SPMS with active disease; SPMS; Secondary Progressive Multiple Sclerosis; siponimod; Mayzent
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — siponimod

INTERVENTIONS:
Drug: Siponimod — 1 or 2 mg film-coated tablets. The tablets have to be taken orally once daily and swallowed whole with water, with or without food.
  Other Names: Mayzent

SUMMARY:
The purpose of this MAP Cohort Treatment Plan is to allow access to siponimod for eligible patients diagnosed with Secondary Progressive Multiple Sclerosis with active disease.

The patient's Treating Physician should follow the suggested treatment guidelines and comply with all local health authority regulations.

The requesting Treating Physician should submit a request for access to the drug (often referred to as Compassionate Use) to Novartis which will be reviewed and assessed by the medical team experienced with the drug and indication.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this Treatment Plan have to meet all of the following criteria:

1. Adult patients who are able to provide written informed consent and have done so Note: proof of efficacy in the Phase III EXPAND study (Kappos et al 2018) has been obtained in patients who were aged 18 to 61 years (inclusive) at screening
2. Diagnosis of SPMS with active disease. The SPMS diagnosis must follow an initial relapsing-remitting disease course of multiple sclerosis (MS) and align with the diagnostic criteria published (Lublin and Reingold 1996, Rovaris et al 2006, Lublin et al 2014)
3. Patient is ambulatory, i.e., has an EDSS score of ≤6.5
4. Patient has no comparable or satisfactory alternative therapy available for treatment of SPMS Written patient informed consent must be obtained prior to start of treatment. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.

Exclusion Criteria:

Patients eligible for this Treatment Plan must not meet any of the following criteria:

1. Disease exclusions

   1. Relapsing-remitting multiple sclerosis
   2. Primary progressive multiple sclerosis
   3. Secondary progressive multiple sclerosis without active disease
2. Medical conditions precluding inclusion such as lab abnormalities or underlying diseases

   1. Patients with an active or stable but treated chronic disease of the immune system other than MS (e.g. rheumatoid arthritis, scleroderma, Sjogren's syndrome, Crohn's disease, ulcerative colitis, etc.) or with a known immunodeficiency syndrome (AIDS, hereditary immune deficiency, drug-induced immune deficiency)
   2. Severe active infections Patients affected by severe infections should only be included after full resolution of the condition
   3. Second-degree AV block Mobitz type II or higher, sick-sinus syndrome, sino-atrial heart block or significant QT prolongation (QTc ≥500 msec).
   4. History of cardiac arrest, recurrent syncope, symptomatic bradycardia, severe cerebrovascular disease, uncontrolled hypertension or severe untreated sleep apnea.
   5. Significant liver disease
   6. Ongoing macular edema (patients with a history of resolved macular edema are allowed to enter the program)
   7. Patients homozygous for CYP2C9*3 (CYP2C9*3*3 genotype)
   8. Patients without a health-care professional confirmed history of chickenpox or documentation of a full course of vaccination with varicella vaccine. They have to undergo antibody testing to varicella zoster virus (VZV) before initiating treatment with siponimod. A full course of vaccination for antibody-negative patients with varicella vaccine is required prior to commencing treatment with siponimod. Initiation of treatment with siponimod has be postponed for one month after completion of the vaccination course to allow full effect of vaccination to occur.
   9. History of hypersensitivity to any drugs or metabolites of similar chemical classes as siponimod.
3. Prior therapy precluding enrollment:

   1. Natalizumab, immunosuppressive/chemotherapeutic medications (e.g. azathioprine, methotrexate) within 6 months prior to enrollment
   2. Rituximab, ofatumumab, ocrelizumab, cladribine, or cyclophosphamide within one year prior to enrollment
   3. Any mitoxantrone during previous two years prior to enrollment or evidence of cardiotoxicity following mitoxantrone or a cumulative life-time dose of more than 60 mg/m2
   4. alemtuzumab, lymphoid irradiation, bone marrow transplantation or other immunosuppressive treatments with effects potentially lasting over 6 months, at any time
4. Concomitant therapy precluding enrollment:

   1. Alemtuzumab, azathioprine, cyclophosphamide, cyclosporine, methotrexate, mitoxantrone, natalizumab, rituximab, ofatumumab, or ocrelizumab as immunosuppressive or immune-modulating therapies
   2. Only during treatment initiation: Class Ia (e.g. quinidine, procainamide), Class III anti-arrhythmic drugs (e.g. amiodarone, sotalol) during treatment initiation
5. Have any of the following out-of-range laboratory values:

   1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST), or gamma-glutamyl transferase (GGT) greater than 5 times the upper limit of normal (ULN) range
   2. White blood cell (WBC) count < 3,500/mm3 (< 3.5 x 109/L)
   3. Lymphocyte count < 800/mm3 (< 0.8 x 109/L)
   4. Serum potassium > ULN
6. Participation in a prior investigational study within 30 days prior to enrollment or within five half-lives of the investigational study drug or until the expected pharmacodynamic effect has returned to baseline, whichever is longer
7. Pregnancy statements and contraception requirements

   1. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
   2. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, UNLESS they are:

      * Women whose partners have been sterilized by vasectomy or other means.
      * Using a highly effective method of birth control for the duration of treatment with siponimod and for at least ten days after stopping treatment with siponimod. Highly effective method of birth control are such resulting in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices (IUDs); periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable.
      * Total abstinence from female-male intercourse (when this is in line with the preferred and usual lifestyle of the subject, if accepted by local regulation)
8. Not able to understand and to comply with treatment instructions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals